CLINICAL TRIAL: NCT03109847
Title: Pilot Study of Metformin to Mitigate Sequelae of Radioactive Iodine Treatment for Well-Differentiated Thyroid Cancers
Brief Title: Metformin to Mitigate Sequelae of Radioactive Iodine Treatment for Thyroid Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16D.564; JT 9411 (Other: JeffTrial Number)
Record Dates: First submitted 2017-03-06; First posted 2017-04-12 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride PO daily for 3 days and then PO BID for up to 2 weeks after completing radioactive iodine treatment.
  Interventions: Drug: Metformin Hydrochloride; Other: Radioactive Iodine
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO daily for 3 days and then PO BID for up to 2 weeks after completing radioactive iodine treatment
  Interventions: Other: Radioactive Iodine; Other: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride — Given Orally
  Other Names: 1,1-Dimethylbiguanide Hydrochloride; 1115-70-4; 91485; Cidophage; Dimefor; Glucoformin; Metformin HCl
  Arms: Arm I (metformin hydrochloride)
Other: Radioactive Iodine — Undergo radioactive iodine treatment
Other: Placebo — Given orally
  Arms: Arm II (placebo)

SUMMARY:
This pilot clinical trial studies how will metformin hydrochloride works in mitigating the side effects of radioactive iodine treatment in patients with differentiated thyroid cancer. Metformin hydrochloride may reduce the metabolic activity of cancer cell and of surrounding supportive tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if treatment with metformin hydrochloride (metformin) inhibits radioactive iodine (RAI)-induced myelosuppression and induces faster recovery of white blood cell count to baseline values, the blood counts will be compared in the pre- and post-treatment samples.

SECONDARY OBJECTIVES:

I. Assess safety and tolerability of metformin treatment in subjects undergoing RAI treatment for differentiated thyroid cancer.

II. To assess the effect of metformin treatment on symptoms of xerostomia, xerophthalmia and dysgeusia as assessed by the Xerostomia Questionnaire (XQ), the modified Vanderbilt Head and Neck Cancer Symposium Survey (version 2.0), University of Washington Quality of Life Questionnaire, and European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTCQLQ)-Head and Neck (H&N)35.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of differentiated thyroid cancer who have undergone total or near-total thyroidectomy and are candidates for iodine I-131 (I-131) treatment at Thomas Jefferson University Hospital (TJUH) are eligible to participate
* Subjects must be diagnosed with differentiated thyroid cancer
* Patients must have previously undergone or plan to undergo thyroidectomy; for those patients who have previously undergone surgery, pre-operative labs, including complete blood cell count with differential must be available
* Patients who have a negative urine pregnancy test prior to enrollment. This should be done as part of pre-admission testing prior to surgery (within 14 days of study enrollment).
* All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Subjects who are pregnant or may become pregnant during metformin administration in accordance with radioactive iodine treatment guidelines
* Subjects on metformin for any reason during the preceding 4 weeks
* Diabetic subjects are eligible if they are not taking metformin, insulin or sulfonylureas
* Subjects who have received iodinated contrast dye. Metformin treatment can be started the day after subjects complete iodinated contrast treatment. If a CT scan with contrast is scheduled after screening and consent, the metformin treatment should be stopped the day before iodinated contrast administration. Metformin can be resumed on the day after last iodinated contrast was administered to the subject.
* Patients with history of hepatic dysfunction or hepatic disease and abnormal liver function tests (previously documented alanine aminotransferase greater than 40 IU/dL and/or plasma aspartate aminotransferase greater than 45 IU/d); patients who have a history of hepatic dysfunction or hepatic disease but whose most recent liver function tests have been documented as normal will be eligible to participate
* Patients with plasma creatinine level greater than 1.3 mg/dL
* Patients with plasma alkaline phosphatase greater than 190 IU/dL
* Patients with plasma bicarbonate less than 22 mEq/L or history of lactic or any other metabolic acidosis
* Patients with history of congestive heart failure
* Patients with myocardial ischemia or peripheral muscle ischemia
* Patients with sepsis or severe infection
* Patients with history of lung disease currently requiring any pharmacologic or supplemental oxygen treatment
* Patients with a current history (in the past 30 days) of heavy drinking which is defined in accordance with CDC definition as more than 8 drinks per week for women and more than 15 drinks per week for men. A standard drink contains .6 ounces of pure alcohol. Generally, this amount of pure alcohol is found in 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor (e.g., gin, rum, vodka, or whiskey). While on study, patients should limit their alcohol consumption to no more than 8 drinks per week for women and no more than 15 drinks per week for men. Patients who feel they cannot comply with this recommendation are not eligible.
* Patients with a systemic disease that could affect their bone marrow or peripheral blood cells (e.g. systemic lupus erythematosus, human immunodeficiency virus infection, rheumatoid arthritis)
* Patients who have received or will receive medication that could affect their hematologic state (tyrosine kinase inhibitors, cytotoxic chemotherapy)
* Patients who are Non-English speaking *Note: This is due to the nature of the study and the process for full translations of the study documents.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Curry, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Started | 6 | 7
Completed | 5 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Red Blood Cell Count From Pre-Resection to Post-Resection
Description: Change in red blood cell count measured from baseline to two weeks after completion of RAI, measured via standard CBC laboratory testing. Longitudinal measures of CBC will be modeled using mixed effects linear regression. Will use a linear contrast to test the null hypothesis that change from pre-resection to post-resection is the same in the control and metformin groups.
Time Frame: Up to 36 months of study duration, an average of 1.5 months
Population: Participants with both pre- and post-treatment CBC values were included in the analysis. Due to missing laboratory data, 4 participants in Arm 1 (Metformin) and 3 participants in Arm 2 (Placebo) were analyzable for this outcome.
Measure: Mean (95% Confidence Interval); unit: million cells per microliter
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Number analyzed (Participants) | 4 | 3
million cells per microliter | -0.11 [-0.74 to 0.51] | -0.63 [-2.70 to 1.45]
Statistical Analysis 1: Comparison: Arm I (metformin hydrochloride) vs Arm II (placebo); Test type: Other; p = 0.404, t-test, 2 sided; Mean Difference (Net) = 0.52, 95% CI 2-sided [-1.26 to 2.29]

2. Primary Outcome: Serum and Salivary Exosome Profile
Description: Will be modeled using mixed effects linear regression
Time Frame: Up to 36 months of study duration
Population: The study terminated early due to poor accrual; no samples collected for exosome profiling. Therefore, no participants were analyzed for this outcome. Data were not collected and the outcome cannot be reported.
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Adverse Events
Description: Number of adverse events assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version v 4.0, from treatment initiation through 15 days post-treatment follow-up.
Time Frame: Up to 36 months of study duration, an average of 1.5 months
Measure: Number; unit: Adverse Events
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Number analyzed (Participants) | 5 | 6
Adverse Events | 32 | 11

4. Secondary Outcome: Xerostomia Assessed by Modified Vanderbilt Head and Neck Cancer Symposium Survey (Version 2.0)
Time Frame: Up to 36 months of study duration
Population: The study terminated early due to poor accrual; no surveys collected for Xerostomia. Therefore, no participants were analyzed for this outcome. Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Xerophthalmia Assessed by Modified Vanderbilt Head and Neck Cancer Symposium Survey (Version 2.0)
Time Frame: Up to 36 months of study duration
Population: The study terminated early due to poor accrual; no surveys collected for Xerophthalmia. Therefore, no participants were analyzed for this outcome. Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Dysgeusia Assessed by Modified Vanderbilt Head and Neck Cancer Symposium Survey (Version 2.0)
Time Frame: Up to 36 months of study duration
Population: The study terminated early due to poor accrual; no surveys collected for Dysgeusia. Therefore, no participants were analyzed for this outcome. Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study period during which adverse events must be reported is normally defined as the period from the initiation of any study procedures to the end of the study treatment follow-up. For this study, the study treatment follow-up is defined as 15 days following the last administration of study treatment, an average of 1.5 months.
Arm/Group | Arm I (metformin hydrochloride) | Arm II (placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 5/6 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (metformin hydrochloride) (N=6) | Arm II (placebo) (N=7)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blurry Vision - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Constipation - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhea - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea - Grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia - Grade 2 (Nervous system disorders) | 1 (1) | 0 (0)
Ear Pain - Grade 1 (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Face Edema - Grade 1 (General disorders) | 0 (0) | 1 (1)
Fatigue - Grade 1 (General disorders) | 1 (2) | 0 (0)
Generalized muscle weakness - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Knee & Achilles Pain - grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea - Grade 1 (Gastrointestinal disorders) | 4 (5) | 0 (0)
Nausea - Grade 2 (Gastrointestinal disorders) | 3 (4) | 1 (1)
Neck Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Upset stomach - Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting - Grade 1 (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting - Grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jaw Pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Numbness - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Sore Throat - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
superficial thrombophlebitis - Grade 2 (Vascular disorders) | 0 (0) | 1 (1)
Weakness - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Xerostomia - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03109847/Prot_SAP_000.pdf